CLINICAL TRIAL: NCT03725878
Title: Effectiveness of Comprehensive Tertiary Interventions on Incidence and Clinical Outcomes of Birth Defects : a Cluster Randomisation Intervention Trial
Brief Title: Effectiveness of Comprehensive Tertiary Interventions on Incidence and Clinical Outcomes of Birth Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Minhang Maternal and Children Health Hospital (Unknown); Songjiang Maternal and Children Health Hospital (Unknown)
Responsible Party: Principal Investigator, Guoying huang, Professor, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016YFC1000500(6)
Record Dates: First submitted 2018-10-24; First posted 2018-10-31 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Birth Defects
Keywords: Birth Defects; periconception; randomized controlled trial; folate
MeSH Terms: conditions — Congenital Abnormalities | interventions — Prenatal Care; Postnatal Care

STUDY DESIGN:
Intervention Model Description: cluster rondomization with average cluster size =100 pregnancies.
Who Masked: Participant
Masking Description: This is a single-blind randomized controlled trial, participants are blinded from their preconceptional folate nutrition status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Standard tertiary interventions of birth defects; Additional preconception health care; Additional health care procedures during and after pregnancy.
  Interventions: Procedure: Standard tertiary interventions of birth defects; Procedure: Additional preconception health care; Procedure: Additional health care procedures during and after pregnancy
- Control (Active Comparator): Standard tertiary interventions of birth defects; Additional health care procedures during and after pregnancy.
  Interventions: Procedure: Standard tertiary interventions of birth defects; Procedure: Additional health care procedures during and after pregnancy

INTERVENTIONS:
Procedure: Standard tertiary interventions of birth defects — Couples eligible for reproductive policy are entitled to routine health cares including general health cares (health education, medical history inquiry, physical examinations, consulting guidance and pregnancy outcome follow-up) and medical examinations (laboratory examinations, virus screenings and image examinations). But nutrients status are not included in these examinations, such as folate, vitamin B12, and macroelements, et al. Regular antenatal cares are required, such as deformity screening by ultrasound. Routine neonatal screenings are conducted to diagnose infant with birth defect timely.
  Other Names: Routine preconception and pregnant health cares
Procedure: Additional preconception health care — Various studies have revealed that folate is essential in early embryo development, whereas folate level evaluation in periconception women is not included in routine health cares. Therefore, we evaluate subject's folate level by serum and red blood cell folate examination. By combination of folate supplement obtained by questionnaire,folate level evaluated by examinations and folate metabolism ability evaluated by genotyping key enzymes in folate metabolism, an individualized folic acid supplementary guide is given to subjects. Red blood cell folate concentration >400 ng/ml before pregnancy is recommended.
  Other Names: Individualized guide for folic acid supplementary
  Arms: Interventional
Procedure: Additional health care procedures during and after pregnancy — Fetus with birth defect will be referred to a tertiary hospital to receive genetic assessments and prenatal diagnosis to reduce unnecessary abortions. A 6-months follow up will be conducted to follow children's birth outcomes. It also helps clinical team to give early diagnosis and treatment for children with birth defect to reduce disability and improve life quality of defect children.
  Other Names: Green channels for antenatal care and postnatal care

SUMMARY:
This project is a single blind cluster randomized controlled trial with a purpose of assessing the effectiveness of a comprehensive tertiary interventions (before pregnancy, during pregnancy and after delivery) on the incidence and the clinical outcomes of birth defects in a preparing-for-pregancy population in Shanghai. The preconception intervention is focused on identifying individuals whose red blood cell folate level is below recommended level for preventing neural tube defects (400ng/ml) or with elevated homocysteine level (over th 80th percentiles, 6.8 µmol/L) , and modifying their folate deficiency status to normal before pregnancy.

DETAILED DESCRIPTION:
According to World health Organization (WHO), approximately 3.2 million children are born with birth defect(s) worldwide and the incidence of birth defects in China is 5.6%. Birth defects are the main cause of fetal death, infant mortality and morbidity, and long-term disability. Congenital heart defects, oral clefts, hydrocephalus, neural tube defects and mental retardation are most common birth defects in China. Though the etiology of birth defects is still unknow, many studies indicated that maternal key nutrition factors, especially maternal folic acid status, during periconception played an important role in organogenesis, reducing the incidence of neural tube defects, congenital heart diseases and some other birth defects.

Our project is a single-blind, cluster randomized controlled trial that aim at evaluating whether hospital-based tertiary intervention approaches reduce the incidence of birth defects (compound primary outcomes, including neural tube defects, congenital heart defects, cleft lips and palates, hydrocephalus, alimentary tract malformations or urological deformities) that identified at middle of gestation via ultrasound or clinical observation at birth. Every couple attending premarital check or preconception physical examination from Minhang and Songjiang district in Shanghai will be recruited. Recruited couples are to draw blood samples and invite to complete questionnaires that collecting informations on diet supplementation. Comprehensive interventions before conception are based on serum folate, red blood cell folate, homocysteine, vitamin B12 and fasting glycemic and lipids profiles. Single nucleotide polymorphisms related to folate and homocysteine matalism pathway will be genotyped in participants with sufficient intake of folic acid but unknown deficiency of the nutrients. Venous blood of pregnant women and questionnaires about the supplementation of key nutrients at the first antenatal visit are also obtained. NT examination, Down's screening, and ultrasound examination results are collected during the second trimester (15-24 gestational week), then routine prenatal genetic counseling, assessment, and diagnosis are provided according to the local policy to those pregnant women with positive screen results indicating high risk of fatal birth defects. Newborns with above mentioned birth defects are provided green channel to clinical specialty team for further diagnosis, surgical correction and rehabilitation guidance. Clinical follow up will be conducted till 6-month old for the prognosis of treatment. The current project will provide evidence on the necessity and effectiveness of preconception intervention focusing on sufficient folate nutrition levels in prevention of birth defects.

ELIGIBILITY:
Inclusion Criteria:

* Females and their husbands attend pre-pregnancy physical examinations from Minhang distrit and Songjiang distrit in Shanghai.
* Couples who have planned to be pregnant within a year
* Women are between 18 and 45 years old

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4808 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Incidence of total fetal birth defects found during the second trimester, still birth, and neontal birth defects identified after delivery | From the confirmation of pregnant to 28 days after birth
  This is a composite outcome: the total number of fetus defects detected by Down's syndrome screenings, NT examinations and Ultrasound image examinations during the second trimester, stillbirth, and the number of birth defects after delivery diagnosed by clinical team.
  (Defects are classified in consistent with our birth defect monitoring policy, which have 24 types of defects: Anencephalus; Spina bifida; Encephalocele; Congenital Hydrocephalus; Cleft Palate; Cleft Lip; Cleft Lip with Cleft Palate; Microtia (including Anotia); Deformity of external ear(s) (except Microtia and Anotia); Esophageal atresia or stenosis; Anorectal atresia (including Congenital Anorectal Malformations); Hypospadia; Ectopocystis; Pes Equinovarus; Polydactylism; Syndactylia; Limb shortening; Congenital Diaphragmatic Hernia; Pcromphalus; Celoschisis; Conjoined Twins; Trisomy 21 syndrome; Congenital heart disease; Others. )

SECONDARY OUTCOMES:
Incidence rate of total abortion because of the affected congenital defects | From the confirmation of pregnant to the 28th gestational week
  Reasons of abortion are recorded
Incidence of death or severe organ dysfunctions | From birth to 6 months after delivery ( can be expanding to the end of the 7th month)
  Severe organ dysfunctions were defined based on specialty clinical examinaitons
Extra medical cost that relates to affecting any birth defects during pregnancy and after birth | From confirmation of pregnancy to one year old after birth
  Additional medical cost that exceeds normal pregnancies and children within one year old
incidence of congenital heart defect | from conception to one year old
  congenital heart defects diagnosed during pregnancy (ultrasound) and after birth( Echocardiography). (Definition see Zhao et al. Lancet 2014)
Total pregnancy loss | from conception to 28 gestational weeks
  artificial abortions without any medical reasons were exluded

CONTACTS AND LOCATIONS:
Overall Officials: Ying G Huang, MD, Ph.D, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu S, Joseph KS, Luo W, Leon JA, Lisonkova S, Van den Hof M, Evans J, Lim K, Little J, Sauve R, Kramer MS; Canadian Perinatal Surveillance System (Public Health Agency of Canada). Effect of Folic Acid Food Fortification in Canada on Congenital Heart Disease Subtypes. Circulation. 2016 Aug 30;134(9):647-55. doi: 10.1161/CIRCULATIONAHA.116.022126. PMID 27572879
- [Background] Czeizel AE, Dudas I, Vereczkey A, Banhidy F. Folate deficiency and folic acid supplementation: the prevention of neural-tube defects and congenital heart defects. Nutrients. 2013 Nov 21;5(11):4760-75. doi: 10.3390/nu5114760. PMID 24284617
- [Background] Ebadifar A, KhorramKhorshid HR, Kamali K, Salehi Zeinabadi M, Khoshbakht T, Ameli N. Maternal Supplementary Folate Intake, Methylenetetrahydrofolate Reductase (MTHFR) C677T and A1298C Polymorphisms and the Risk of Orofacial Cleft in Iranian Children. Avicenna J Med Biotechnol. 2015 Apr-Jun;7(2):80-4. PMID 26140186
- [Derived] Li M, Zhang Y, Chen X, Wang D, Ji M, Jiang Y, Dou Y, Ma X, Sheng W, Yan W, Huang G. Effectiveness of community-based folate-oriented tertiary interventions on incidence of fetus and birth defects: a protocol for a single-blind cluster randomized controlled trial. BMC Pregnancy Childbirth. 2020 Aug 20;20(1):475. doi: 10.1186/s12884-020-03154-w. PMID 32819312

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03725878/SAP_001.pdf